CLINICAL TRIAL: NCT04435106
Title: Compassionate Use of Opaganib in Patients With Severe COVID-19
Brief Title: Compassionate Use of Opaganib in Patients With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0123-20- SZMC
Record Dates: First submitted 2020-05-26; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infections
MeSH Terms: conditions — Coronavirus Infections | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide; Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Opaganib + Standard of Care: Study participants received opaganib 2 x 250 mg capsules (500 mg) every 12 hours in addition to Standard of Care
  Interventions: Drug: Opaganib; Drug: Standard of Care
- Standard of Care: Study participants received Standard of Care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Opaganib — Study participants received opaganib 2 x 250 mg capsules (500 mg) every 12 hours in addition to Standard of Care
  Other Names: Yeliva; ABC294640
  Groups: Opaganib + Standard of Care
Drug: Standard of Care — Study participants received Standard of Care

SUMMARY:
Shaare-Zedek Medical Center is a tertiary academic hospital in Jerusalem, Israel. On March 2020, a dramatic increase in the number of COVID-19 cases were diagnosed in Jerusalem. RedHill Biopharma, Ltd. offered opaganib under compassionate use for the treatment of COVID-19 patients. Eligible patients were those hospitalized with COVID-19 confirmed by a reverse-transcriptase-polymerase-chain-reaction assay. Patients received opaganib and Standard of Care. For the purpose of this study, the opaganib and Standard of Care patient group was compared to a group of patients that received only Standard of Care. Opaganib is an investigational drug under development and not approved for commercial distribution.

DETAILED DESCRIPTION:
In this observational study, the two cohorts were assigned retrospectively. Patients either received opaganib and Standard of Care (SOC) or SOC only. All patients were defined by the treating physicians at baseline as severe COVID-19. For the control cohort, IRB approval was granted to collect de-identified data. Both cohorts had similar median age and similar rates of diabetes, hypertension and obesity.

The two treatment groups, opaganib and SOC vs. SOC were then analyzed for their clinical outcomes including baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with COVID-19 confirmed by a reverse-transcriptase-polymerase-chain-reaction assay
* patients with severe disease requiring oxygen support via high-flow nasal cannula
* signed informed consent
* acceptable liver and renal function tests
* acceptable hematologic status

Exclusion Criteria:

* pregnant or nursing women
* patients on warfarin, apixaban, argatroban or rivaroxaban
* patients with New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe COVID-19 who required oxygen support via high-flow nasal cannula (HFNC)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Measure the time to weaning from high-flow nasal cannula | Every day from day 1 to day 14
Measure the time to breathing ambient (room) air | Every day from day 1 to day 14

SECONDARY OUTCOMES:
Measure change in lymphocyte count | On day of admission or day 1 of treatment and every 2-4 days, till day 14
Measure change in C-reactive protein | On day of admission or day 1 of treatment and every 2-4 days, till day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare-Zedek Medical Center, Jerusalem, Israel